CLINICAL TRIAL: NCT03392571
Title: Phase II Multi-Center Study of Nab-paclitaxel, Gemcitabine and Cisplatin (NGC-Triple Regimen as Preoperative Therapy in Patients With Potentially Resectable and Borderline Resectable Pancreatic Cancer
Brief Title: Phase II Study of NGC-Triple Regimen in Potentially Resectable Pancreatic Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped due to lack of funding
Sponsor: Pancreatic Cancer Research Team (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCRT 17-001
Record Dates: First submitted 2017-12-06; First posted 2018-01-08 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Resectable Pancreatic Cancer
Keywords: Resectable pancreatic cancer, NGC-triple regimen
MeSH Terms: interventions — Gemcitabine; Cisplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Patients receive 3 cycles of preoperative chemotherapy. The regimen consists of gemcitabine 800 mg/m2, nab-paclitaxel 100 mg/m2 and cisplatin 25 mg/m2 given IV weekly x 2, every 3 weeks (one cycle).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Resectable and borderline restable (Experimental): Potentially operable or borderline resectable pancreatic adenocarcinoma as assessed by standard CT criteria and histologically confirmed.
  Patients receive 3 cycles of preoperative chemotherapy (NGC-triple regimen). The regimen consists of gemcitabine 800 mg/m2, Nab-paclitaxel 100 mg/m2and Cisplatin 25 mg/m2 given IV weekly x 2, every 3 weeks (one cycle).
  Patients will be evaluated for adjuvant therapy within 12 weeks of surgery which will consist of Nab-paclitaxel, gemcitabine, and Cisplatin IV weekly x 2, every 3 weeks (one cycle) x 3 cycles.
  Interventions: Drug: NGC-Triple regimen

INTERVENTIONS:
Drug: NGC-Triple regimen — gemcitabine 800 mg/m2; Abraxane (nab-paclitaxel 100 mg/m2; cisplatin 25 mg/m2
  Other Names: gemcitabine; cisplatin; Nab-paclitaxel

SUMMARY:
This is a phase II multi-center study of nab-paclitaxel, gemcitabine and cisplatin (NGC triple regimen) as preoperative therapy in potentially resectable pancreatic cancer patients.

DISEASE STATE

* Potentially operable or borderline resectable pancreatic adenocarcinoma as assessed by standard CT criteria and histologically confirmed.
* Staging by pancreatic protocol, helical abdominal computed tomography (with contrast) or MRI (with contrast) required (endoscopic ultrasound is not required).
* No evidence of metastatic disease. Lymphadenopathy (defined as nodes measuring >1 cm in short axis) outside the surgical basin (i.e., para-aortic, peri-caval, celiac axis, or distant nodes) is considered M1 (unless nodes are biopsied and are negative, then enrollment can be considered after review with the study PI).

Potentially Resectable Pancreatic Cancer

* No involvement of the celiac artery, common hepatic artery, and superior mesenteric artery (SMA) and, if present, replaced right hepatic artery.
* No involvement or <180° interface between tumor and vessel wall of the portal vein and/or superior mesenteric vein (SMV-PV) and patent portal vein/splenic vein confluence.
* For tumors of the body and tail of the pancreas, involvement of the splenic artery and vein of any degree is considered resectable disease. Borderline Resectable Pancreatic Cancer
* Tumor-vessel interface ≥180° of vessel wall circumference, and/or reconstructible occlusion of the SMV-PV.
* Tumor-vessel interface <180° of the circumference of the SMA.
* Tumor-vessel interface <180° of the circumference of the celiac artery.
* Reconstructible short-segment interface of any degree between tumor and hepatic artery.

DETAILED DESCRIPTION:
The purpose of this study is to find out if the study drugs nab-paclitaxel, cisplatin, and gemcitabine given together are safe and effective. The combination of nab-paclitaxel plus gemcitabine has been studied in treating patients with pancreatic cancer, and as of September, 2013 is approved for the treatment of advanced pancreatic cancer. In this study, cisplatin will be added to nab-paclitaxel plus gemcitabine, and tested in people who have not yet had any cancer therapy for the diagnosis of localized pancreatic cancer, as treatment prior to surgery, with the goal of improving response.

Another name for nab-paclitaxel is Abraxane®. Nab-paclitaxel contains the same medication as the prescription chemotherapy drug Abraxane®. Nab-paclitaxel is approved by the FDA for the treatment of advanced breast cancer, and in September, 2013 nab-paclitaxel, combined with gemcitabine, was approved by the FDA for the treatment of advanced pancreatic cancer.

Cisplatin is approved by the FDA for the treatment of advanced bladder cancer, advanced ovarian cancer, and advanced testicular cancer and other childhood cancers. However, cisplatin is not approved by the FDA for the treatment of advanced pancreatic cancer.

Gemcitabine was approved by the FDA in 1996 for the treatment of pancreatic cancer. It is also an approved treatment for ovarian cancer, lung cancer, and breast cancer.

Nab-paclitaxel, cisplatin, and gemcitabine will be given weekly for 2 weeks followed by a week of rest, for a total of 3 cycles. A cycle is defined as one set of 3 weeks of chemotherapy treatment. Patients will undergo surgery after a minimum of 3 weeks after Cycle 3 of chemotherapy. Following surgery, patients mayl be treated for up to 3 cycles of this same chemotherapy combination.

ELIGIBILITY:
Major Inclusion Criteria for the Study Include the Following:

* Patient has an ECOG performance status PS 0-1. No prior chemotherapy or radiation for pancreatic cancer and no prior exposure to gemcitabine and/or nab-paclitaxel

Patient has the following blood counts at baseline:

* ANC ≥1.5 × 109/L (1500 /mm3)
* Platelets ≥100 × 109/L; (100,000/mm3)
* Hgb ≥10 g/dL

Patient has the following blood chemistry levels at baseline:

* AST (SGOT), ALT (SGPT) ≤ 3.0 × upper limit of normal (ULN)
* Alkaline phosphatase (AP) ≤3.0 X ULN
* Total bilirubin ≤1.5 or ≤ULN
* Serum creatinine ≤1.5mg/dL or calculated clearance ≥50 mL/min/1.73 m2 for patients with serum creatinine levels >1.5 mg/dL
* Patient has acceptable coagulation status as indicated by a PT within normal limits (± 15%) and PTT within normal limits (± 15%)

Major Exclusion Criteria include the Following:

1. Patient has locally advanced unresectable pancreatic cancer.
2. Patients aged >75.
3. Histologies other than adenocarcinoma, or any mixed histologies, will NOT be eligible.
4. Patient uses therapeutic Coumadin for a history of pulmonary emboli or DVT.
5. Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
6. Patient has known infection with HIV, hepatitis B, or hepatitis C.
7. Patient has undergone major surgery, other than diagnostic surgery (i.e. surgery done to obtain a biopsy for diagnosis without removal of an organ) within 4 weeks prior to Day 1 of treatment in this study.
8. Prior chemotherapy or radiation for pancreatic cancer. Prior exposure to gemcitabine and/or nab-paclitaxel.
9. Patient has a history of allergy or hypersensitivity to the study drugs.

   -

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate 2 year survival from date of entry into study | Patients will be followed for survival from Day 1 of treatment with phone calls or review of records on a monthly basis for the first 6 months, and then every 6 months for 24 months.
  Overall survival of patients as well as 1, and 2 year survivals will be tabulated.

SECONDARY OUTCOMES:
Determine the number and type of treatment-related adverse events as assessed by CTCAE 4.0 | Monitor treatment-related adverse events during neoadjuvant treatment for up to 3 months prior to surgery, and for up to 3 months after surgery.
  To determine the number and type of treatment-related adverse events as assessed by CTCAE v4.0
Histological Response to Pre-Operative Therapy | Specimens obtained during surgery 3-7 weeks following last dose of chemotherapy;
  Grade III/IV histological response to preoperative therapy in resected tumor specimens
Radiological Response Rate to Pre-Operative Therapy in the Primary Tumor | PET/CT scans performed at Baseline, and immediately prior to surgery, 3-7 weeks following last dose of chemotherapy;
  Radiological response rate in the primary tumor to preoperative therapy
CA 19-9 response to preoperative therapy | CA 19-9 evaluation during preoperative therapy once per treatment cycle;
  CA 19-9 response to preoperative therapy
Resectability (RO and R1) Rate Following Preoperative Therapy | Determine RO and R1 resectability rate at surgery, 3-7 weeks following last dose of chemotherapy;
  Resectability (RO and R1) rate following preoperative therapy in potentially operable or locally advanced patients
Determine Postoperative Complications of Surgery | Evaluate surgical complications within 12 weeks post-surgery to determine eligibility for up to 3 cycles (28 days per cycle) of adjuvant treatment
  Tabulate postoperative complications of surgery
Time to Recurrence | After Day 1 of treatment, time to recurrence will be collected within the 24 month follow up period
  Determine Time to recurrence and patterns of recurrence within the 24 month follow-up period